CLINICAL TRIAL: NCT07057336
Title: Evaluation of Post-Operative Pain Following the Use of Nano-Calcium Hydroxide as an Intracanal Medicament: A Randomized Controlled Trial
Brief Title: Evaluation of Post-Operative Pain Following the Use of Nano-Calcium Hydroxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Büşra Över Kılıç, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 05.04.2024/143
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Chronic Apical Periodontitis
Keywords: Calcium Hydroxide; Nanocalcium Hydroxide; Postoperative pain; Chronic apical periodontitis; Intracanal medicament
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Calcium Hydroxide (CH) (Experimental): Following completion of canal shaping with rotary instrumentation and irrigation using 5 mL of 2.5% sodium hypochlorite (NaOCl), canals were flushed sequentially with 5 mL distilled water, 5 mL of 17% ethylenediaminetetraacetic acid (EDTA), another 5 mL of distilled water, 5 mL of 2.5% NaOCl, and finally 5 mL of distilled water. Canals were then dried using sterile paper points. Conventional calcium hydroxide (CH) paste was introduced into the canal using a Lentulo spiral. A sterile cotton pellet was placed in the pulp chamber, and the cavity was sealed with glass ionomer cement.
  Interventions: Drug: Conventional Calcium Hydroxide (CH)
- Nanocalcium Hydroxide (NCH) (Experimental): Following completion of canal shaping with rotary instrumentation and irrigation using 5 mL of 2.5% sodium hypochlorite (NaOCl), canals were flushed sequentially with 5 mL distilled water, 5 mL of 17% ethylenediaminetetraacetic acid (EDTA), another 5 mL of distilled water, 5 mL of 2.5% NaOCl, and finally 5 mL of distilled water. Canals were then dried using sterile paper points. Nanocalcium hydroxide (NCH) paste was placed into the canal using a Lentulo spiral to ensure uniform distribution. The access cavity was temporarily restored with a sterile cotton pellet and glass ionomer cement.
  Interventions: Drug: Nanocalcium Hydroxide (NCH)

INTERVENTIONS:
Drug: Conventional Calcium Hydroxide (CH) — Following completion of canal shaping with rotary instrumentation and irrigation using 5 mL of 2.5% sodium hypochlorite (NaOCl), canals were flushed sequentially with 5 mL distilled water, 5 mL of 17% ethylenediaminetetraacetic acid (EDTA), another 5 mL of distilled water, 5 mL of 2.5% NaOCl, and finally 5 mL of distilled water. The cavity was sealed temporarily with a sterile cotton pellet and glass ionomer cement. Conventional calcium hydroxide was retained for 7 days before final obturation.
  Arms: Conventional Calcium Hydroxide (CH)
Drug: Nanocalcium Hydroxide (NCH) — Following completion of canal shaping with rotary instrumentation and irrigation using 5 mL of 2.5% sodium hypochlorite (NaOCl), canals were flushed sequentially with 5 mL distilled water, 5 mL of 17% ethylenediaminetetraacetic acid (EDTA), another 5 mL of distilled water, 5 mL of 2.5% NaOCl, and finally 5 mL of distilled water. The cavity was sealed temporarily with a sterile cotton pellet and glass ionomer cement. Nanocalcium hydroxide was retained for 7 days before final obturation.
  Arms: Nanocalcium Hydroxide (NCH)

SUMMARY:
The goal of this clinical trial is to evaluate the effect of different intracanal medicaments-conventional calcium hydroxide (CH) and nano-sized calcium hydroxide (NCH)-on the intensity of postoperative pain following root canal treatment in asymptomatic necrotic single-rooted teeth.

The primary research question of this study is as follows:

Does the use of nano-sized calcium hydroxide, compared to conventional calcium hydroxide, result in significantly reduced postoperative pain after root canal treatment?

In both groups, standardized instrumentation will be performed using rotary NiTi files and 2.5% sodium hypochlorite irrigation. After cleaning and shaping, canals will be medicated with either CH or NCH, followed by temporary sealing.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Single-rooted permanent maxillary or mandibular teeth
* Asymptomatic teeth with necrotic pulps confirmed by negative response to cold test
* Presence of periapical radiolucency (PAI score 2-5)
* No sensitivity to percussion or palpation
* Patients who signed informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Systemic diseases requiring antibiotic prophylaxis (e.g., infective endocarditis, immunosuppression)
* Use of antibiotics, corticosteroids, or analgesics within the past 7 days
* History of chemotherapy or radiotherapy
* Uncontrolled diabetes mellitus or hypertension
* Chronic renal failure, hematologic disorders
* Teeth with root resorption, previous endodontic treatment, or multirooted anatomy
* Teeth with periodontal pockets >4 mm or mobility
* Inability to attend follow-up visits
* Patients with extensive coronal destruction rendering definitive restoration unfeasible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | up to 72 hours
  The visual analog scale for pain is a straight line with one end meaning no pain (0) and the other end meaning the worst pain (10) imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. It may be used to help choose the right dose of pain medicine. Also called VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdi Oğuz Yoldaş, DDS PHD, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amir N, Mansoor E, Eeman N, Ahmed MN, Mansoor E, Mansoor E, Hussain K, Afreixo V, Mansoor A, Brochado Martins JF, Palma PJ. Jasminum-based Nano-reinforced Calcium Hydroxide Reduces Postoperative Pain in Symptomatic Apical Periodontitis: A Randomized Controlled Trial. J Endod. 2025 Aug;51(8):996-1005. doi: 10.1016/j.joen.2025.05.016. Epub 2025 Jun 2. PMID 40466913